CLINICAL TRIAL: NCT05539326
Title: A Multicenter, Single- Arm Postmarket Study of the Construct Validity of Community Walking Speed Data Collected Remotely With the Canary canturioTM te Tibial Extension
Brief Title: A Study of the Construct Validity of Community Walking Speed Data Collected Remotely With the Canary canturioTM te Tibial Extension
Status: Completed | Type: Observational
Sponsor: Canary Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: POS-CTE-002P
Record Dates: First submitted 2022-09-10; First posted 2022-09-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis, Knee
Keywords: total knee arthroplasty; Canary canturio™te with Canary Health Implanted Reporting Processor; clinical outcomes; 4 meter walk test
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PIQ Patients: Patient is scheduled for or has undergone primary total knee arthroplasty (TKA) using a Persona Personalized Knee System with Canary Tibial Extension (PIQ) TKA implant according to the appropriate surgical technique and IFU. If you decide to take part in this research study, the general procedures include one follow-up visit where you will be asked to complete two performance-based tests that are used to assess your physical function following Total Knee Arthroplasty ("TKA"). As part of your standard of care, you will receive a Zimmer Persona® Personalized Knee System with Canary canturioTM (CTE) tibial extension. As part of this study, subjects will be asked to perform two performance based tests called the 4 meter walk test and the timed up and go test. Subjects will also be asked to complete a series of patient questionnaires that will assess their post-operative function.
  Interventions: Other: Performance Clinical Outcome Test

INTERVENTIONS:
Other: Performance Clinical Outcome Test — Patients will be asked to perform a fast 4-meter walk test (4mWT) and the Timed up and Go (TUG) test in the clinic during their post-operative follow-up visit. Both performance exams will be performed in a controlled environment within the physician's clinic.

SUMMARY:
The purpose of this study is to determine the construct validity of the Canary Tibial Extension's measure of self-selected community walking speed. Construct validity will be assessed by the Pearson's correlation coefficient between self-selected community walking speed and the 4-meter walk test. The objective of this multicenter, prospective study is to demonstrate that remote measurement of community walking speed with the Canary canturioTM (CTE) tibial extension is correlated with the fast 4-meter walk test (4mWT).

DETAILED DESCRIPTION:
The primary endpoint is community walking speed, calculated as a mean, remotely captured over the 7 days prior to the patient's regularly scheduled office visit: specifically, the correlation (Pearson correlation coefficient) of community walking speed with the 4mWT.

The secondary endpoints are as follows:

* Correlation coefficient between community walking speed and the Timed Up and Go (TUG) Test
* Completeness of data collection and transmission by the study device
* Correlation coefficient between community walking speed and the Oxford Knee Score
* Correlation coefficient between community walking speed and the Knee Injury and Osteoarthritis Outcome Score Jr (KOOS JR)

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older at the time of surgery
* Patient is scheduled for or has undergone primary total knee arthroplasty using a Persona Personalized Knee System with Canary Tibial Extension (PIQ) TKA implant according to the appropriate surgical technique and IFU.
* Patient must be willing and able to complete the protocol required follow-up
* Patient has participated in the study-related informed consent process
* Patient has a platform-compatible personal computer located in their dwelling with substantially reliable wireless internet access and a USB port

Exclusion Criteria:

* Simultaneous bilateral TKA
* Staged bilateral TKA less than 6 months from indexed procedure
* Patient is a current alcohol or drug abuser
* Patient is known to be pregnant, breastfeeding, or considered a member of a protected class (e.g., prisoner, mentally incompetent, etc.)
* Patient has a psychiatric illness or cognitive deficit that will not allow proper informed consent and participation in follow-up program
* Patient has previous history of infection in the affected joint and/or a local or systemic infection that may affect the prosthetic joint
* Patient with mental or neurologic conditions who are unwilling or incapable of following postoperative care instructions
* Patient with Neuropathic Arthropathy
* Patient has rheumatoid arthritis accompanied by an ulcer of the skin or a history of recurrent breakdown of the skin
* Patient is undergoing procedures or treatments using ionizing radiation
* Patient has a known or suspected sensitivity to one or more of the implant materials.
* Patients with known orthopaedic lower extremity, spinal and/or neurologic conditions that could affect gait

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient is scheduled for or has undergone primary total knee arthroplasty using a Persona Personalized Knee System with Canary Tibial Extension (PIQ) TKA implant according to the appropriate surgical technique and IFU.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
4 Meter Walk Test | 4 wks+2 weeks post TKA
  A 4MWT test will be performed in the physician's clinic along a clear pathway of at least 8 in length in a designated area over solid flooring. The 8-m distance will be measured with a starting (0m) and an end point (8m) with additional marks at 2m and 6m to identify the 4m which is the timed portion of the test. A handheld, calibrated stopwatch will be used as the gold standard for measuring walking speed output during the 4 mWT, measuring the time it takes to complete the test.
Timed Up and Go Test *(TUG) | 4 wks+2 weeks post TKA
  Patients may use a walking aid if needed. Patients will begin by sitting back in a standard armchair. Investigator will identify a line 3 meters (9.8 feet) away on the floor. When the investigator says "go" the patient will:
  1. stand up from the chair
  2. walk to the line on the floor at a comfortable and safe walking speed
  3. turn and walk back to the chair at a comfortable and safe walking speed
  4. Sit down again A stopwatch will be used to record the time it takes from the initiation of the exam on the word "go" to the end of the exam when the patient's buttocks touch the seat.
Community Walking Speed | 7 days prior to follow-up appoinment
  Average walking speed

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | wks+2 weeks post TKA
  Patient Reported Outcome on level of Pain
Oxford Knee Score | wks+2 weeks post TKA
  Patient Reported Outcome on Clinical Function
KOOS Jr | 4wks+2 weeks post TKA
  Patient Reported Outcome on Clinical Function
Clinical Limping Evaluation | 4wks+2 weeks post TKA
  Self Evaluation of Limping

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Vail Summit Orthopaedics and Neurosurgery, Frisco, Colorado
  - South Bend Orthopaedics, South Bend, Indiana
  - Mississippi Sports Medicine and Orthopaedic Center, Jackson, Mississippi
  - Orthopedic NJ, Sparta, New Jersey
  - Dr. Ballard, Oregon City, Oregon
  - Orthopaedic Surgery and Sports Medicine, San Antonio, Texas